CLINICAL TRIAL: NCT04994548
Title: Endoscopic Resection of Early Esophageal Tumors in the Context of Cirrhosis or Portal Hypertension: a Multicenter Observational Study
Brief Title: Endoscopic Resection of Early Esophageal Tumors in the Context of Cirrhosis or Portal Hypertension
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2019PI67
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Esophageal Neoplasms; Cirrhosis; Portal Hypertension
MeSH Terms: conditions — Esophageal Neoplasms; Fibrosis; Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cirrhotic patients or with portal hypertension: Patients with early esophageal cancer
  Interventions: Procedure: Endosocpic resection of early esophageal tumor

INTERVENTIONS:
Procedure: Endosocpic resection of early esophageal tumor — under general anesthesia, by mucosectomy or endoscopic submucosal dissection

SUMMARY:
Cirrhotic patients may be at high risk for esophageal cancer. Endoscopic resection is the standard treatment for superficial tumors. However, cirrhosis might be associated with upper gastrointestinal bleeding, particularly in case of portal hypertension or coagulopathy. This study aims to assess safety, efficacy and methods to prevent potential complications in cirrhosis or portal hypertension context for esophageal endoscopic resection.

This retrospective multicentric French-Belgian study includes all consecutive patients with cirrhosis or portal hypertension who underwent esophageal endoscopic resection from January 2005 to 2021.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years with cirrhosis or portal hypertension who underwent endoscopic resection of an early esophageal tumor

Exclusion Criteria:

* younger than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 112 patients with cirrhosis or portal hypertension who underwent endoscopic resection of an early esophageal tumor
Enrollment: 112 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2005-02-03 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
technical success of early esophageal cancer resection | baseline
  defined by a complete macroscopic resection

SECONDARY OUTCOMES:
adverse events per procedure (immediate bleeding, perforation) | baseline
morbidity post procedure (delayed bleeding, infection, esophageal stenosis, 30-days related liver decompensation, 30-days related mortality) | up to 4 weeks
Potential risk factors for adverse events | baseline
preemptive methods to the risk of bleeding | baseline

IPD SHARING:
Plan to Share IPD: No